CLINICAL TRIAL: NCT02723201
Title: A Randomized, Open Label Phase 1 Study in Healthy Volunteers to Evaluate the Relative Bioavailability of a Single Dose of Various Test Solid Formulations of TAK-020 Compared With a Single Dose of Reference Oral Solution and to Evaluate the Food Effect and Potentially the Dose Proportionality of the Optimal Solid Dose Formulation
Brief Title: TAK-020 Relative Bioavailability and Food Effect Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-020-1002; U1111-1171-4650 (Registry Identifier: WHO); 2015-002635-18 (EudraCT Number); 16/WA/0012 (Registry Identifier: NRES)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part-1, Period 1: TAK-020 17.5 mg Oral Solution (Experimental): Single dose 17.5 milligram (mg), on Day 1, followed by 7 days of washout. Dose will be determined from TAK-020 single rising dose (SRD) trial.
  Interventions: Drug: TAK-020 Captisol Oral Solution
- Part-1, Period 2: TAK-020 17.5 mg Co-crystal Tablet (CCT) (Experimental): Single oral dose 17.5 mg, on Day 1, followed by 7 days of washout. Dose will be the same as Part 1, Period 1.
  Interventions: Drug: TAK-020 CCT
- Part-1, Period 3:TAK-020 17.5 mg Solid Dispersion Tablet (SDT) (Experimental): Single oral dose 17.5 mg, on Day 1, followed by 7 days of washout. Dose will be the same as Part 1, Period 1.
  Interventions: Drug: TAK-020 SDT
- Part-1, Period 4:TAK-020 17.5 mg Immediate Release Tablet(IRT) (Experimental): Single oral dose 17.5 mg, on Day 1, followed by 7 days of washout. Dose will be the same as Part 1, Period 1.
  Interventions: Drug: TAK-020 IRT
- Part 2, Period 1: TAK-020 25 mg CCT (Experimental): Participants will be randomized to AB or BA crossover where A= Fasted, B =Fed. Sequence I: Single oral dose TAK-020 25 mg, Fasted (A), 7 days washout, single oral dose TAK-020 Fed (B) Sequence II: Single oral dose TAK-020 25 mg, Fed (B), 7 days washout, single oral dose TAK-020 Fasted (A) Dose will be determined from SRD trial and Part 1.
  Interventions: Drug: TAK-020 CCT
- Part- 3 Cohort 1: TAK-020 Solid Formulation (Experimental): Single oral dose on Day 1. Dose will be determined from SRD trial and Parts 1 and 2
  Interventions: Drug: TAK-020 Solid Formulation
- Part 3 Cohort 2: TAK-020 Solid Formulation (Experimental): Single oral dose on Day 1. Dose will be determined from SRD trial and Parts 1 and 2
  Interventions: Drug: TAK-020 Solid Formulation

INTERVENTIONS:
Drug: TAK-020 Captisol Oral Solution — TAK-020 solution.
  Arms: Part-1, Period 1: TAK-020 17.5 mg Oral Solution
Drug: TAK-020 CCT — TAK-020 co-crystal tablet
  Arms: Part-1, Period 2: TAK-020 17.5 mg Co-crystal Tablet (CCT)
Drug: TAK-020 SDT — TAK-020 Solid dispersion tablet.
  Arms: Part-1, Period 3:TAK-020 17.5 mg Solid Dispersion Tablet (SDT)
Drug: TAK-020 IRT — TAK-020 immediate release tablet.
  Arms: Part-1, Period 4:TAK-020 17.5 mg Immediate Release Tablet(IRT)
Drug: TAK-020 CCT — TAK-020 co-crystal tablet.
  Arms: Part 2, Period 1: TAK-020 25 mg CCT
Drug: TAK-020 Solid Formulation — TAK-020 solid formulation
  Arms: Part 3 Cohort 2: TAK-020 Solid Formulation; Part- 3 Cohort 1: TAK-020 Solid Formulation

SUMMARY:
The purpose of this study is to assess the relative bioavailability of solid oral formulations of TAK-020 in comparison with single dose of TAK-020 oral solution formulation and to evaluate the food effect and potentially the dose proportionality of the optimal oral solid formulation.

DETAILED DESCRIPTION:
TAK-020 is being developed for the potential treatment of autoimmune diseases including rheumatoid arthritis. Currently TAK-020 is available as an oral solution. This study is to develop an oral tablet formulation. There are three parts to this study. Part 1 will compare different tablet formulations of TAK-020 compared to a reference oral solution to identify the best tablet formulation to use in Parts 2 and 3. Part 2 will look at the effect food has on TAK-020. Part 3 is optional; its implementation will be decided upon using data from Part 2. It will evaluate whether increased doses of TAK-020 produce an expected proportional increase in the plasma concentration of TAK-020.

In Part 1 participants will receive a single dose of the following:

Period 1: TAK-020 Oral Solution Period 2: TAK-020 Co-Crystal Tablet Period 3: TAK-020 Solid Dispersion Tablet Period 4: TAK-020 Immediate Release Tablet

In Part 2 participants will be split into two groups; one will receive the chosen formulation of TAK-020 in the fasted state followed by the fed state and the other group will receive it in the fed state followed by the fasted state. The dose used in Part 2 will be based upon data from Part 1 and previous studies.

Participants in Part 3 of the study will be split into 2 cohorts. Each cohort will be administered, in the fasted state, a single dose of the tablet selected as optimal from previous study parts. The dose used will be based upon data from Parts 1 and 2 and previous studies.

Part 1 will assess the relative bioavailability of TAK-020 by using analysis of variance (ANOVA) on tmax, and the natural logarithms of AUCs, and Cmax. Part 2 will assess the food effect of TAK-020, also using ANOVA on tmax, and the natural logarithms of AUCs, and Cmax. The power model will be used to assess dose proportionality of single doses of the solid formulations in the fasted state from Parts 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. Is legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy adult male or female.
4. Is aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
5. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) between 18 and 32 kilogram per square meter (kg/m^2), inclusive at Screening and Day -1.
6. Male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose of study medication.
7. Female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent and throughout the duration of the study and until the next menstrual period or 90 days after exit from the study, whichever is first. If the next menstrual period is delayed, a pregnancy test will be required for exclusion of pregnancy.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Has a known hypersensitivity to any component of the formulation of TAK-020, Captisol, or related compounds.
4. Has a positive urine drug result for drugs of abuse or a positive breath alcohol screen at Screening or Check-in (Day -1).
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as 4 or more alcoholic units per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
6. Has taken any excluded medication, supplements, or food products listed in Prohibited Medications and Foods table.
7. If female, is pregnant or lactating or intending to become pregnant before, during or within 3 months after exit from this study (90 days post last dose); or intending to donate ova during such time period.
8. If male, the participant intends to donate sperm during the course of this study or for 90 days after the last dose of study drug.
9. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash.
10. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [example, cholecystectomy]).
11. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
12. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
13. Has poor peripheral venous access.
14. Has donated or lost 450 mililiter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
15. Has a Screening or Check-in (Day -1) abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or medically qualified subinvestigator.
16. Has QT interval with Fridericia correction method (QTcF) greater than (>) 430 millisecond (msec) for men and >450 msec for women or PR outside the range of 120 to 220 msec confirmed upon repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
17. Has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities:

    1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.2* the upper limit of normal (ULN).
    2. Positive screen test for drugs of abuse.
    3. Positive blood screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus-1 or -2 antibodies (test done at Screening visit only).
    4. A positive test for tuberculosis (TB) (QuantiFERON) (test done at Screening Visit only).
18. Vaccination with any live vaccine within 4 weeks of study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-28; Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 28 April 2016 to 24 August 2016.
Pre-assignment Details: Healthy participants were enrolled in 3 part study to receive TAK-020. Part-1: relative bio-availability of solid formulations, Part-2: effect of food on co-crystal tablet(CCT) and Part-3: dose linearity of CCT. Part-3 was not conducted, as relative bioavailability of solid formulation was greater than(>) 50% compared with oral solution of TAK-020.
Groups:
- Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT: TAK-020 17.5 milligram (mg), oral solution (OS), under fasted state, once on Day 1 of first intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, CCT, orally, under fasted state, once on Day 1 of second intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, solid dispersion tablets (SDT), orally, under fasted state, once on Day 1 of third intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, immediate release tablets (IRT), orally, under fasted state, once on Day 1 of fourth intervention period.
- Part 2- TAK-020 25 mg CCT: Fasted + Fed: TAK-020 25 mg, CCT, orally, under fasted state, once on Day 1 of first intervention period, followed by 7 days of washout period, further followed by TAK-020 25 mg, CCT, orally, under fed, once on Day 1 of second intervention period.
- Part 2- TAK-020 25 mg CCT: Fed + Fasted: TAK-020 25 mg, CCT, orally, under fed state, once on Day 1 of first intervention period, followed by 7 days of washout period, further followed by TAK-020 25 mg, CCT, orally, under fasted state, once on Day 1 of second intervention period.
Period: First Intervention Period
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 11 | 7 | 7
Completed | 11 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 11 | 7 | 7
Completed | 11 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 11 | 7 | 7
Completed | 9 | 7 | 7
Not Completed | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Washout Period 2
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Part 1- TAK-020 17.5 mg: OS + CCT + SDT + IRT | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Groups:
- Part 1: TAK-020 17.5 mg: TAK-020 17.5 mg, OS, under fasted state, once on Day 1 of first intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, CCT, orally, under fasted state, once on Day 1 of second intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, SDT, orally, under fasted state, once on Day 1 of third intervention period; followed by 7 days washout period, followed by TAK-020 17.5 mg, IRT, orally, under fasted state, once on Day 1 of fourth intervention period.
- Total: Total of all reporting groups
Arm/Group | Part 1: TAK-020 17.5 mg | Part 2- TAK-020 25 mg CCT: Fasted + Fed | Part 2- TAK-020 25 mg CCT: Fed + Fasted | Total
Number analyzed (Participants) | 11 | 7 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (8.82) | 31.1 (6.49) | 38.9 (12.36) | 39.3 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 7 | 4 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 7 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 7 | 7 | 24
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 11 | 7 | 7 | 25
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.7 (10.40) | 172.3 (7.36) | 173.0 (6.51) | 172.2 (8.34)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 78.16 (16.448) | 74.26 (11.454) | 75.50 (10.207) | 76.32 (13.212)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.23 (3.140) | 24.91 (2.724) | 25.19 (2.884) | 25.57 (2.900)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 10 | 6 | 5 | 21
  Current smoker | 0 | 0 | 0 | 0
  Ex-smoker | 1 | 1 | 2 | 4
Alcohol Classification [Count of Participants; unit: Participants]
  Never drinks | 0 | 1 | 0 | 1
  Current drinker | 10 | 6 | 6 | 22
  Ex-drinker | 1 | 0 | 1 | 2
Caffeine/Xanthine Classification [Count of Participants; unit: Participants]
  Caffeine/xanthine consumption | 10 | 7 | 7 | 24
  No caffeine/xanthine consumption | 1 | 0 | 0 | 1
Female Reproductive Status [Count of Participants; unit: Participants]
  Surgically sterile | 3 | 1 | 0 | 4
  Female of childbearing potential | 1 | 2 | 1 | 4
  Not applicable (male participants) | 7 | 4 | 6 | 17
Amount of Alcohol Consumed by Participant [Count of Participants; unit: Participants] — Population: Baseline measure was analyzed only for those participants who were current drinker and had alcohol consumption.
  Participants
    number analyzed (Participants) | 10 | 6 | 6 | 22
    Less than (<) 4 drinks per day | 10 | 6 | 6 | 22
    4 or more drinks per day | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-020
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The pharmacokinetic (PK) set where Day 1 assessment were available. The PK set included all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part 1: TAK-020 17.5 mg OS: TAK-020 17.5 mg, OS, once under fasted state on Day 1 of first intervention period. A washout period of 7 day was maintained between each intervention period.
- Part 1: TAK-020 17.5 mg CCT: TAK-020 17.5 mg, CCT, orally under fasted state, once on Day 1 of second intervention period. A washout period of 7 day was maintained between each intervention period.
- Part 1: TAK-020 17.5 mg SDT: TAK-020 17.5 mg, SDT, orally under fasted state, once on Day 1 of third intervention period. A washout period of 7 day was maintained between each intervention period.
- Part 1: TAK-020 17.5 mg IRT: TAK-020 17.5 mg, IRT, orally under fasted state, once on Day 1 of fourth intervention period.
- Part 2: TAK-020 25 mg CCT Fasted: TAK-020 25 mg, CCT, orally under fasted state, once on Day 1 of either first intervention period or second intervention period.
- Part 2: TAK-020 25 mg CCT Fed: TAK-020 25 mg, CCT, orally under fed state, once on Day 1 of either first intervention period or second intervention period.
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
nanogram per milliliter (ng/mL) | 104.182 (35.0658) | 44.800 (26.4189) | 139.522 (71.6739) | 6.012 (1.8606) | 63.314 (34.1699) | 40.629 (17.6750)
Statistical Analysis 1: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg CCT; Analysis of variance (ANOVA) was performed on the natural logarithms of Cmax with regimen as the fixed effects and participant as the random effect. The point estimate and 90 percent (%) confidence interval (CI) was obtained by taking the antilog of the difference in the log transformed least square (LS) means and its CI, respectively; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.402, 90% CI 2-sided [0.320 to 0.505]
Statistical Analysis 2: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg SDT; ANOVA was performed on the natural logarithms of Cmax with regimen as the fixed effects and participant as the random effect. The point estimate and 90% CI was obtained by taking the antilog of the difference in the log transformed LS means and its CI, respectively; Test type: Superiority or Other; p = 0.249, ANOVA; LS Mean Difference = 1.216, 90% CI 2-sided [1.016 to 1.455]
Statistical Analysis 3: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg IRT; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.055, 90% CI 2-sided [0.041 to 0.074]
Statistical Analysis 4: Comparison: Part 2: TAK-020 25 mg CCT Fasted vs Part 2: TAK-020 25 mg CCT Fed; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.054, ANOVA; LS Mean Difference = 0.685, 90% CI 2-sided [0.499 to 0.939]

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-020
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set where Day 1 assessment were available. The PK set included all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
hour | 0.530 [0.50 to 1.00] | 1.000 [0.50 to 2.00] | 0.750 [0.50 to 1.00] | 1.000 [0.75 to 6.00] | 1.000 [0.50 to 2.00] | 2.000 [0.75 to 4.03]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-020
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 10 | 9 | 8 | 13 | 13
nanogram*hour per milliliter (ng*hr/mL) | 257.455 (97.5416) | 164.485 (72.4927) | 316.448 (127.4409) | 32.783 (18.5993) | 220.396 (89.7255) | 185.935 (29.6651)
Statistical Analysis 1: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg CCT; ANOVA was performed on the natural logarithms of AUC∞ with regimen as the fixed effects and participant as the random effect. The point estimate and 90% CI was obtained by taking the antilog of the difference in the log transformed LS means and its CI, respectively; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean Difference = 0.648, 90% CI 2-sided [0.497 to 0.844]
Statistical Analysis 2: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg SDT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.423, ANOVA; LS Mean Difference = 1.180, 90% CI 2-sided [1.088 to 1.279]
Statistical Analysis 3: Comparison: Part 1: TAK-020 17.5 mg OS vs Part 1: TAK-020 17.5 mg IRT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean Difference = 0.116, 90% CI 2-sided [0.077 to 0.176]
Statistical Analysis 4: Comparison: Part 2: TAK-020 25 mg CCT Fasted vs Part 2: TAK-020 25 mg CCT Fed; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.037, ANOVA; LS Mean Difference = 0.836, 90% CI 2-sided [0.731 to 0.957]

4. Primary Outcome: Terminal Disposition Phase Half-life (T1/2z) in Plasma for TAK-020
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 10 | 9 | 8 | 13 | 13
hour | 4.695 (1.0781) [0.50 to 1.00] | 4.661 (1.4147) [0.50 to 2.00] | 3.976 (0.9787) [0.50 to 1.00] | 5.005 (2.8545) [0.75 to 6.00] | 6.183 (0.8914) [0.50 to 2.00] | 4.412 (1.2323) [0.75 to 4.03]

5. Secondary Outcome: Number of Participants Who Experience at Least One or More Treatment-emergent Adverse Event (TEAE)
Time Frame: Baseline up to 30 days after last dose of study drug (Day 58 in Part 1), (Day 40 in Part 2)
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
participants | 1 | 3 | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants Who Meet the Takeda Markedly Abnormal Criteria for Clinical Laboratory Tests at Least Once Post Dose
Time Frame: Baseline up to Day 2
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
participants
  Hematology | 1 | 0 | 0 | 0 | 0 | 0
  Chemistry | 0 | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Meet the Takeda Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Time Frame: Baseline up to Day 2
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
participants | 0 | 1 | 2 | 2 | 6 | 5

8. Secondary Outcome: Number of Participants Who Meet the Takeda Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Baseline up to Day 2
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Number analyzed (Participants) | 11 | 11 | 9 | 9 | 14 | 14
participants | 5 | 5 | 4 | 4 | 5 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and up to 30 days after last dose of study drug (Day 58 in Part 1), (Day 40 in Part 2)
Description: At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings.Any event spontaneously reported by participant/observed by investigator was recorded,irrespective of relation to study treatment.Number at risk included those participants who have actually received the mentioned intervention during study.
Arm/Group | Part 1: TAK-020 17.5 mg OS | Part 1: TAK-020 17.5 mg CCT | Part 1: TAK-020 17.5 mg SDT | Part 1: TAK-020 17.5 mg IRT | Part 2: TAK-020 25 mg CCT Fasted | Part 2: TAK-020 25 mg CCT Fed
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/9 | 0/9 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/11 | 3/11 | 0/9 | 0/9 | 1/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: TAK-020 17.5 mg OS (N=11) | Part 1: TAK-020 17.5 mg CCT (N=11) | Part 1: TAK-020 17.5 mg SDT (N=9) | Part 1: TAK-020 17.5 mg IRT (N=9) | Part 2: TAK-020 25 mg CCT Fasted (N=14) | Part 2: TAK-020 25 mg CCT Fed (N=14)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.